CLINICAL TRIAL: NCT06273735
Title: Evaluation of Intra- and Postoperative Cardiac Events in Patients With Localised Prostate Carcinoma and Radical Prostatectomy
Brief Title: Prospective Trial: Acute Myocardial Injury After Radical Prostatectomy
Status: Completed | Type: Observational
Sponsor: Martini-Klinik am UKE GmbH (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-PS-33b; PV7350 (Other: Martini-Klinik)
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Myocardial Injury
Keywords: acute myocardial injury; Myocardial Injury after Noncardiac Surgery; radical prostatectomy; prostate cancer; complication; Clavien-Dindo; Myocardial infarction; Revised Cardiac Risk Index
MeSH Terms: conditions — Prostatic Neoplasms; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- radical prostatectomy patients with versus without acute myocardial injury: The cohort consists of open and robotic-assisted radical prostatectomy patients. The rate of acute myocardial injury is determined by laboratory chemistry as part of the study as well as clinically through routine visits and postoperatively through questionnaires. Intervention is not performed according to the study protocol but is part of the normal clinical course, if necessary.
  Interventions: Diagnostic Test: Pre- and postoperative determination of troponin as part of the study and 24-month FU survey

INTERVENTIONS:
Diagnostic Test: Pre- and postoperative determination of troponin as part of the study and 24-month FU survey — An intervention is carried out as part of the normal clinical procedure regardless of the study measurement parameters.

SUMMARY:
This prospective observational study investigates the incidence of acute myocardial injury after radical prostatectomy for prostate cancer. Consecutive patients undergoing elective open or robot-assisted radical prostatectomy at the Martini-Klinik are included. High-sensitivity cardiac troponin I (hs-cTnI) is measured preoperatively and on postoperative days 1 and 2 to identify acute myocardial injury, defined according to the 4th Universal Definition of Myocardial Infarction. Secondary outcomes include the incidence of myocardial infarction, major adverse cardiac and cerebrovascular events, and mortality during the hospital stay and at 24 months. Baseline patient characteristics (age, BMI, cardiovascular risk factors including the Revised Cardiac Risk Index, comorbidities, and prior cardiac therapy) as well as surgical and tumor-specific parameters are recorded. Associations between acute myocardial injury and clinical variables are analyzed.

DETAILED DESCRIPTION:
Primary endpoint:

Acute myocardial injury, defined as a postoperative troponin concentration above the 99th percentile sex-specific upper reference limit with a) an increase of ≥ 50% from baseline if the baseline troponin I or T concentration was below the 99th percentile sex-specific upper reference limit or with b) an increase of ≥ 20% from baseline if the baseline troponin I or T concentration was above the 99th percentile sex-specific upper reference limit. percentile or with b) an increase of ≥ 20 % compared to the initial value if the initial troponin I or T concentration was above the sex-specific upper reference limit of the 99th percentile.

Secondary endpoints:

1. recording the frequency of acute myocardial damage without or with clinical findings typical of ischaemia.
2. frequency of cardiovascular events during hospitalisation. Cardiovascular events are defined as follows: non-fatal cardiac arrest, heart failure, interventional coronary angiography, coronary artery bypass surgery, new-onset atrial fibrillation, stroke, pulmonary artery embolism, deep vein thrombosis of leg or arm.
3. correlation between the level of postoperative troponin increase and the occurrence of cardiovascular events during hospitalisation.
4. predictive value of the Revised Cardiac Risk Index for the occurrence of acute myocardial damage.
5. differences in the incidence of acute myocardial damage in open radical prostatectomies versus minimally invasive radical prostatectomies.

Furthermore, the included patients are followed up for 24 months and questioned about cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Consent form signed
* Patients with a biopsy-proven prostate carcinoma
* planned ORP or RARP

Exclusion Criteria:

* No exclusion of patients who fulfil the above inclusion criteria

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with biopsy-proven prostate cancer who undergo open or robotic-assisted radical prostatectomy at the Martini Clinic are included (N=1000).
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
rate of acute myocardial injury in standardised open and robot-assisted radical prostatectomy | the day before surgery until 24months follow-up
  Survey of the rate of asymptomatic and symptomatic myocardial damage. A troponin determination is carried out before the prostatectomy as well as a troponin determination on the first and second postoperative day. An ACS is recorded clinically. Myocardial events and treatment of myocardial infarction are also recorded during the follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Graefen, Prof., Study Director — Martini-Klinik am UKE GmbH
Locations (1):
- Martini-Klinik am UKE GmbH, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
A publication in a peer-reviewed journal is planned.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: First publications are planned for 2024.
Access Criteria: A publication in a peer-reviewed journal is planned.

REFERENCES:
- [Background] Pearse RM, Moreno RP, Bauer P, Pelosi P, Metnitz P, Spies C, Vallet B, Vincent JL, Hoeft A, Rhodes A; European Surgical Outcomes Study (EuSOS) group for the Trials groups of the European Society of Intensive Care Medicine and the European Society of Anaesthesiology. Mortality after surgery in Europe: a 7 day cohort study. Lancet. 2012 Sep 22;380(9847):1059-65. doi: 10.1016/S0140-6736(12)61148-9. PMID 22998715
- [Background] Smilowitz NR, Gupta N, Guo Y, Berger JS, Bangalore S. Perioperative acute myocardial infarction associated with non-cardiac surgery. Eur Heart J. 2017 Aug 14;38(31):2409-2417. doi: 10.1093/eurheartj/ehx313. PMID 28821166
- [Background] Botto F, Alonso-Coello P, Chan MT, Villar JC, Xavier D, Srinathan S, Guyatt G, Cruz P, Graham M, Wang CY, Berwanger O, Pearse RM, Biccard BM, Abraham V, Malaga G, Hillis GS, Rodseth RN, Cook D, Polanczyk CA, Szczeklik W, Sessler DI, Sheth T, Ackland GL, Leuwer M, Garg AX, Lemanach Y, Pettit S, Heels-Ansdell D, Luratibuse G, Walsh M, Sapsford R, Schunemann HJ, Kurz A, Thomas S, Mrkobrada M, Thabane L, Gerstein H, Paniagua P, Nagele P, Raina P, Yusuf S, Devereaux PJ, Devereaux PJ, Sessler DI, Walsh M, Guyatt G, McQueen MJ, Bhandari M, Cook D, Bosch J, Buckley N, Yusuf S, Chow CK, Hillis GS, Halliwell R, Li S, Lee VW, Mooney J, Polanczyk CA, Furtado MV, Berwanger O, Suzumura E, Santucci E, Leite K, Santo JA, Jardim CA, Cavalcanti AB, Guimaraes HP, Jacka MJ, Graham M, McAlister F, McMurtry S, Townsend D, Pannu N, Bagshaw S, Bessissow A, Bhandari M, Duceppe E, Eikelboom J, Ganame J, Hankinson J, Hill S, Jolly S, Lamy A, Ling E, Magloire P, Pare G, Reddy D, Szalay D, Tittley J, Weitz J, Whitlock R, Darvish-Kazim S, Debeer J, Kavsak P, Kearon C, Mizera R, O'Donnell M, McQueen M, Pinthus J, Ribas S, Simunovic M, Tandon V, Vanhelder T, Winemaker M, Gerstein H, McDonald S, O'Bryne P, Patel A, Paul J, Punthakee Z, Raymer K, Salehian O, Spencer F, Walter S, Worster A, Adili A, Clase C, Cook D, Crowther M, Douketis J, Gangji A, Jackson P, Lim W, Lovrics P, Mazzadi S, Orovan W, Rudkowski J, Soth M, Tiboni M, Acedillo R, Garg A, Hildebrand A, Lam N, Macneil D, Mrkobrada M, Roshanov PS, Srinathan SK, Ramsey C, John PS, Thorlacius L, Siddiqui FS, Grocott HP, McKay A, Lee TW, Amadeo R, Funk D, McDonald H, Zacharias J, Villar JC, Cortes OL, Chaparro MS, Vasquez S, Castaneda A, Ferreira S, Coriat P, Monneret D, Goarin JP, Esteve CI, Royer C, Daas G, Chan MT, Choi GY, Gin T, Lit LC, Xavier D, Sigamani A, Faruqui A, Dhanpal R, Almeida S, Cherian J, Furruqh S, Abraham V, Afzal L, George P, Mala S, Schunemann H, Muti P, Vizza E, Wang CY, Ong GS, Mansor M, Tan AS, Shariffuddin II, Vasanthan V, Hashim NH, Undok AW, Ki U, Lai HY, Ahmad WA, Razack AH, Malaga G, Valderrama-Victoria V, Loza-Herrera JD, De Los Angeles Lazo M, Rotta-Rotta A, Szczeklik W, Sokolowska B, Musial J, Gorka J, Iwaszczuk P, Kozka M, Chwala M, Raczek M, Mrowiecki T, Kaczmarek B, Biccard B, Cassimjee H, Gopalan D, Kisten T, Mugabi A, Naidoo P, Naidoo R, Rodseth R, Skinner D, Torborg A, Paniagua P, Urrutia G, Maestre ML, Santalo M, Gonzalez R, Font A, Martinez C, Pelaez X, De Antonio M, Villamor JM, Garcia JA, Ferre MJ, Popova E, Alonso-Coello P, Garutti I, Cruz P, Fernandez C, Palencia M, Diaz S, Del Castillo T, Varela A, de Miguel A, Munoz M, Pineiro P, Cusati G, Del Barrio M, Membrillo MJ, Orozco D, Reyes F, Sapsford RJ, Barth J, Scott J, Hall A, Howell S, Lobley M, Woods J, Howard S, Fletcher J, Dewhirst N, Williams C, Rushton A, Welters I, Leuwer M, Pearse R, Ackland G, Khan A, Niebrzegowska E, Benton S, Wragg A, Archbold A, Smith A, McAlees E, Ramballi C, Macdonald N, Januszewska M, Stephens R, Reyes A, Paredes LG, Sultan P, Cain D, Whittle J, Del Arroyo AG, Sessler DI, Kurz A, Sun Z, Finnegan PS, Egan C, Honar H, Shahinyan A, Panjasawatwong K, Fu AY, Wang S, Reineks E, Nagele P, Blood J, Kalin M, Gibson D, Wildes T; Vascular events In noncardiac Surgery patIents cOhort evaluatioN (VISION) Writing Group, on behalf of The Vascular events In noncardiac Surgery patIents cOhort evaluatioN (VISION) Investigators; Appendix 1. The Vascular events In noncardiac Surgery patIents cOhort evaluatioN (VISION) Study Investigators Writing Group; Appendix 2. The Vascular events In noncardiac Surgery patIents cOhort evaluatioN Operations Committee; Vascular events In noncardiac Surgery patIents cOhort evaluatioN VISION Study Investigators. Myocardial injury after noncardiac surgery: a large, international, prospective cohort study establishing diagnostic criteria, characteristics, predictors, and 30-day outcomes. Anesthesiology. 2014 Mar;120(3):564-78. doi: 10.1097/ALN.0000000000000113. PMID 24534856
- [Background] Vascular Events In Noncardiac Surgery Patients Cohort Evaluation (VISION) Study Investigators; Devereaux PJ, Chan MT, Alonso-Coello P, Walsh M, Berwanger O, Villar JC, Wang CY, Garutti RI, Jacka MJ, Sigamani A, Srinathan S, Biccard BM, Chow CK, Abraham V, Tiboni M, Pettit S, Szczeklik W, Lurati Buse G, Botto F, Guyatt G, Heels-Ansdell D, Sessler DI, Thorlund K, Garg AX, Mrkobrada M, Thomas S, Rodseth RN, Pearse RM, Thabane L, McQueen MJ, VanHelder T, Bhandari M, Bosch J, Kurz A, Polanczyk C, Malaga G, Nagele P, Le Manach Y, Leuwer M, Yusuf S. Association between postoperative troponin levels and 30-day mortality among patients undergoing noncardiac surgery. JAMA. 2012 Jun 6;307(21):2295-304. doi: 10.1001/jama.2012.5502. PMID 22706835
- [Background] Puelacher C, Lurati Buse G, Seeberger D, Sazgary L, Marbot S, Lampart A, Espinola J, Kindler C, Hammerer A, Seeberger E, Strebel I, Wildi K, Twerenbold R, du Fay de Lavallaz J, Steiner L, Gurke L, Breidthardt T, Rentsch K, Buser A, Gualandro DM, Osswald S, Mueller C; BASEL-PMI Investigators. Perioperative Myocardial Injury After Noncardiac Surgery: Incidence, Mortality, and Characterization. Circulation. 2018 Mar 20;137(12):1221-1232. doi: 10.1161/CIRCULATIONAHA.117.030114. Epub 2017 Dec 4. PMID 29203498
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). Glob Heart. 2018 Dec;13(4):305-338. doi: 10.1016/j.gheart.2018.08.004. Epub 2018 Aug 25. No abstract available. PMID 30154043